CLINICAL TRIAL: NCT04472962
Title: The Effect of a Low-carbohydrate-high-protein Pre-exercise Meal on Exercise-induced Hypoglycemia in People With Type 1 Diabetes.
Brief Title: The Importance of Meal Composition on Preventing Exercise-induced Hypoglycemia in People With Type 1 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H-20007316
Record Dates: First submitted 2020-06-24; First posted 2020-07-16 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2020-12

CONDITIONS: Type 1 Diabetes
Keywords: Exercise; Nutrition; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-carbohydrate-high-protein pre-exercise meal (Active Comparator)
  Interventions: Other: Pre-exercise meal
- High-carbohydrate-low-protein pre-exercise meal (Active Comparator)
  Interventions: Other: Pre-exercise meal

INTERVENTIONS:
Other: Pre-exercise meal — Mixed meal with low-carbohydrate-high-protein content
  Arms: Low-carbohydrate-high-protein pre-exercise meal
Other: Pre-exercise meal — Mixed meal with high-carbohydrate-low-protein content
  Arms: High-carbohydrate-low-protein pre-exercise meal

SUMMARY:
This study is a clinical, randomized, crossover study. The study investigates the effect of a low-carbohydrate-high-protein pre-exercise meal on preventing exercise-induced hypoglycemia in people with type 1 diabetes. The hypothesis is that intake of a low-carbohydrate-high-protein meal can reduce the duration and depth of hypoglycemia during and after exercise in people with type 1 diabetes compared with an isocaloric high-carbohydrate-low-protein meal with identical fat content. The study will contribute with new knowledge about importance of meal composition on preventing exercise-induced hypoglycemia.

DETAILED DESCRIPTION:
Background:

People with type 1 diabetes practicing a low-carbohydrate diet can increase the fat and/or protein content of the diet to cover their energy needs. In relation to physical activity, ingestion of protein is preferable for muscle protein synthesis and enhances structural changes in non-muscle tissues such as tendons and bones. Furthermore, addition of ≥ 28 g of protein to a meal is likely to result in significant and sustained postprandial hyperglycemia commencing in the late postprandial period (2-3 h) and continuing beyond 5 h in people with type 1 diabetes. The protein-induced change in the postprandial glucose response could be beneficial in relation to prevention of exercise-induced hypoglycemia. Hypoglycemia is a common fear in people with type 1 diabetes and makes many abstain from exercising.

This study investigates the effect of a low-carbohydrate-high-protein pre-exercise meal on preventing exercise-induced hypoglycemia in people with type 1 diabetes. The hypothesis is that intake of a low-carbohydrate-high-protein meal can reduce the duration and depth of hypoglycemia during and after exercise in people with type 1 diabetes compared with an isocaloric high-carbohydrate-low-protein meal with identical fat content.

This study will contribute with new knowledge about importance of meal composition on preventing exercise-induced hypoglycemia. The study may add new aspects to current guidelines for glucose management during exercise in people with type 1 diabetes. If the strategy has a positive effect on preventing exercise-induced hypoglycemia it will be useful to all people with type 1 diabetes irrespective of diet strategy.

Study design:

The study is a randomized, two-arm crossover trial including one screening visit, two study days and a short visit after each study day, where the participants must meet to upload research data. The study will include adults with type 1 diabetes on insulin pump therapy using flash glucose monitoring (FGM) or continuous glucose monitoring (CGM). 15 participants have to complete the study. The study days are identical except for the content of the pre-exercise meal (low-carbohydrate-high-protein meal versus high-carbohydrate-low-protein meal) and the size of the meal bolus. Meals are isocaloric. The participants will complete two study days in random order with a 10-14 days washout period between. 48 hours prior to each study day blood glucose will be monitored by CGM and activity level will be monitored by an activity monitor wristband.

Each study day is divided into an in-clinic period, which takes place at Steno Diabetes Center Copenhagen (SDCC), and a home period, which takes place in the participants own homes.

The participants will arrive at the research facility in the morning following an overnight fast. A pre-exercise meal with either low-carbohydrate-high-protein content or high-carbohydrate-low-protein content will be served. To estimate the gastric emptying 1g paracetamol will be added to the meal. After ingesting the meal and 90 min of resting the participants must perform 45 min of exercise on an ergometer cycle equaling to 60 % of their peak oxygen consumption or until hypoglycemia (plasma glucose < 3.9) or unbearable symptoms of hypoglycemia. Throughout the in-clinic study day the participants must use their insulin pumps. The basal insulin rate and meal-bolus will be adjusted according to international guidelines. Blood samples for analysis of glucose, insulin, glucagon, cortisol, adrenalin, noradrenalin, growth hormone, ketones, lactate, free fatty acids, GLP1, GIP and inflammatory markers will be collected. Indirect calorimetry will be performed before, during and after exercise to measure energy expenditure, respiratory exchange ratio and carbohydrate and fat oxidation rates. The Borg Scale will be used to assess perceived exertion during the exercise and a visual analog scale will be used to assess the feeling of satiety during the study day.

Leaving SDCC the home period begins. Throughout the home period the blood glucose and activity level will be monitored by the CGM and the activity monitor until the next morning, where the study day ends. From the research facility the participants will be provided a standard evening meal and a bedtime snack. The participants will also be provided dextrose tablets, which they must ingest in case of hypoglycemia. Within one week after both study days, the participants must meet at the clinic to upload research data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years.
* Type 1 diabetes ≥ 5 years.
* Insulin pump use ≥ 1 year.
* Use of flash glucose monitoring (FGM) or continuous glucose monitoring (CGM) ≥ 3 months.
* Body mass index 18.5-30 kg/m2.
* HbA1c ≤ 64 mmol/mol (8.0%).
* Self-reported hypoglycemia awareness
* Ability to carbohydrate count for all meals.
* Familiarity with the insulin pump bolus calculator for all meals.
* Moderate to vigorous level of physical activity

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start.
* Use of Metronic Minimed 670G insulin pump system.
* Allergy to paracetamol or nuts
* Females who are pregnant, breast-feeding or intend to become pregnant.
* Heart disease.
* Severe asthma.
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the individual unsuitable for study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
The area over the curve (AOC). | 7 hours.
  The primary outcome measure is the AOC for plasma glucose (PG) < 3.9 mmol/L during the in-clinic period assessed by YSI (Yellow Spring Instruments 2900 STAT Plus). The AOC is the area, which extends from the plasma glucose curve to the limit for hypoglycemia < 3.9 mmol/l.

SECONDARY OUTCOMES:
Time spent < 3.9 mmol/l during in-clinic period, home period and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Time spent < 3.9 mmol/l during in-clinic period assessed by YSI. | 7 hours.
Time spent 3.0-3.8 mmol/l during in-clinic period, home period, and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Time spent 3.0-3.8 mmol/l during in-clinic period assessed by YSI. | 7 hours.
Time spent < 3.0 mmol/l during in-clinic period, home period, and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Time spent < 3.0 mmol/l during in-clinic period assessed by YSI. | 7 hours.
Time spent 3.9-10.0 mmol/l during in-clinic period, home period and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Time spent > 10.0 mmol/l during in-clinic period, home period and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Time spent > 10.0 during in-clinic period assessed by YSI. | 7 hours.
Time spent > 13.9 during in-clinic period, home period and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Time spent > 13.9 during in-clinic period assessed by YSI. | 7 hours.
Glycemic variability (% coefficient of variation) during in-clinic, home, and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Glycemic variability (% coefficient of variation) during in-clinic period assessed by YSI. | 7 hours.
Standard deviation (SD) during in-clinic period, home period, and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Standard deviation (SD) during in-clinic period assessed by YSI. | 7 hours.
Number of hypoglycemia events (< 3.9 mmol/l) in-clinic period, home period and overall study period assessed by CGM. | 7, 17 and 24 hours respectively.
Number of hypoglycemia events (< 3.9 mmol/l) during in-clinic period assessed by YSI. | 7 hours.
Amount of dextrose in grams ingested to treat hypoglycemia (< 3.9 mmol/l) during in-clinic period, home period and overall study period. | 7, 17 and 24 hours respectively.
Peak PG/blood glucose after ingestion of pre-exercise meal assessed by YSI and CGM. | 3 hours
Time-to-peak PG/blood glucose after ingestion of pre-exercise meal assessed by YSI and CGM | 3 hours
Area under the curve of total insulin during in-clinic period | 7 hours
Area under the curve of glucagon during the in-clinic period. | 7 hours
Area under the curve of cortisol during the in-clinic period. | 7 hours
Area under the curve of growth hormone during the in-clinic period. | 7 hours
Area under the curve of epinephrine during the in-clinic period. | 7 hours
Area under the curve of norepinephrine during the in-clinic period. | 7 hours
Area under the curve of lactate during the in-clinic period. | 7 hours
Area under the curve of free fatty acids during the in-clinic period. | 7 hours
Area under the curve of ketones during the in-clinic period. | 7 hours
Area under the curve of GLP-1 during the in-clinic period | 7 hours
Area under the curve of GIP during the in-clinic period | 7 hours
Area under the curve of IL6 during the in-clinic period | 7 hours
Area under the curve of IL-1ra during the in-clinic period | 7 hours
Area under the curve of IL-10 during the in-clinic period | 7 hours
Area under the curve of TNFα during the in-clinic period | 7 hours
Area under the curve of IL-1β during the in-clinic period | 7 hours
Respiratory exchange ratio (RER) during the in-clinic period | 7 hours
Energy expenditure during the in-clinic period (kcal/min) | 7 hours
Carbohydrate and fat oxidation rates during the in-clinic period | 7 hours.
Time of gastric emptying after ingestion of the pre-exercise meal assessed by serum paracetamol. | 7 hours.
Physical performance during the exercise phase evaluated by heart rate | 45 minutes
Physical performance during the exercise phase evaluated by watt | 45 minutes
Feeling of physical hardness during the exercise phase evaluated using the Borg Scale. | 45 minutes.
Satiety (assessed by visual analog scale after pre-exercise meal) during the in-clinic period | 7 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kristensen KB, Ranjan AG, McCarthy OM, Holst JJ, Bracken RM, Norgaard K, Schmidt S. Effects of a Low-Carbohydrate-High-Protein Pre-Exercise Meal in Type 1 Diabetes-a Randomized Crossover Trial. J Clin Endocrinol Metab. 2023 Dec 21;109(1):208-216. doi: 10.1210/clinem/dgad427. PMID 37463489
- [Derived] McCarthy OM, Kristensen KB, Christensen MB, Schmidt S, Ranjan AG, Nicholas C, Bain SC, Norgaard K, Bracken R. Metabolic and physiological responses to graded exercise testing in individuals with type 1 diabetes using insulin pump therapy. Diabetes Obes Metab. 2023 Mar;25(3):878-888. doi: 10.1111/dom.14938. Epub 2023 Jan 3. PMID 36482870